CLINICAL TRIAL: NCT04224064
Title: Identification of a New Blood Biomarker for the Diagnosis and Prognosis of Liposarcomas
Acronym: ESPACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PROICM 2019-09 ESP
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Liposarcoma; Atypical Lipomatous Tumor
Keywords: Liposarcoma; Cancer; Atypical Lipomatous Tumor; New non-invasive biological test
MeSH Terms: conditions — Liposarcoma; Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy subjects cohort (Experimental): A single blood sample will be made in healthy subjects.
  Interventions: Diagnostic Test: Blood sampling
- Liposarcoma patients cohort (Experimental): Blood samples will be collected at different times: one before induction before surgery and then the second 4 weeks after surgery (+/- 1 week), then every 3 months for 18 months.
  Interventions: Diagnostic Test: Blood sampling

INTERVENTIONS:
Diagnostic Test: Blood sampling — Blood samples will be performed in fasted state for the controls and the patients. A single sample will be made in healthy subjects and several samples in patients: one before induction before surgery and then the second 4 weeks after surgery (+/- 1 week), then every 3 months for 18 months.

SUMMARY:
The main objective of this project is to identify a new non-invasive biological test for the diagnosis of LPS by measuring circulating serine levels. The current gold standard is the detection of Mdm2 amplification by the FISH.

DETAILED DESCRIPTION:
Sarcomas are rare diseases, accounting for less than 1% of all malignant diseases in adults¹. Their incidence is about 6 new cases per 100,000 in inhabitants per year, ie 4,000 to 5,000 new cases estimated per year in France.

Liposarcoma (LPS) is the most common soft tissue sarcoma subtype, accounting for approximately 15% of all sarcomas.

The OMS classification distinguishes 5 categories of LPS: myxoid, pleomorphe, round-cell liposarcomas, dedifferentiated (DD-LPS) and well-differentiated (WD-LPS). Research team is interested by the last two in this study.

The diagnosis is suspected on the imaging examinations (MRI for limb tumors and CT for retro-peritoneal LPS) which should lead to a discussion at a multidisciplinary tumor board in an expert center to validate the biopsy for definitive diagnosis and define the best biopsy route to avoid the risk of spread. In France, the management of patients with sarcoma is organized around the network of 24 "NETSARC" centers.

WD-LPS and DD-LPS, may be difficult to distinguish from benign adipose tumors and undifferentiated sarcomas, respectively. Molecular analyze, based on the detection of Mdm2 gene amplification by Fluorescence in situ Hybridization (FISH) is currently the "gold standard". It is performed on a tumor biopsy. The biopsy is a radiologic biopsy as it is recommended in the guidelines to reduce the risk of disease spread. The material allowing the diagnosis is thus limited complicating the realization of morphology, immunohistochemistry and molecular biology on the same sample. The other limitation is that this tumor fragment does not always reflect intra-tumor heterogeneity.

The treatment is surgical with monobloc resection by a surgeon specialized in sarcomas. Despite surgical excision, the risk of local and distant recurrence is approximately 26% for well-differentiated liposarcomas⁵ and up to 59% for dedifferentiated retroperitoneal liposarcomas. Prognostic factors for recurrence are the quality of excision, tumor size, grade, and retroperitoneal / limb localization. The problematic concerning these 2 types of liposarcomas is not the same. In WD-LPS, the question is to know the risk of recurrence in case of unplanned R1 resection (representing approximately 50% of initial surgeries). Indeed a systematic surgical revision of all these cases is expensive and morbid whereas in 50% of cases no tumor residue will be found on the surgical recovery. For the DD-LPS the problem is different because the surgical revision must be systematic in case of non-R0 surgery, but it is the risk of local recurrence despite adequate surgery and the metastatic risk that must be evaluated in order to propose an adjuvant treatment (chemotherapy and / or radiotherapy) to patients with a high risk of recurrence also making it essential to identify a biological factor of prognosis to select patients with a high risk of relapse.

Clinicians propose to identify a new blood test that would indicate the presence of the disease. It would then serve for the diagnosis but also prognosis allowing us to evaluate the residual disease after surgery of excision. Due to the complexity of sarcomas, identifying an effective and reliable biomarker for WD-LPS and DD-LPS with non-invasive methods is a challenge, but clinicians hope that their project will provide a more efficient and patient-friendly method for the detection of the disease. Our project relies on the complementary expertise provided by clinicians, researchers and biostatisticians in close collaboration.

Clinicians have recently characterized a novel function of the p53 independent Mdm2 protein in serine metabolism, which could play a fundamental role in the development of LPS. Through pan-genome approaches clinicians have characterized a novel transcriptional activity of Mdm2 and demonstrated its role in the metabolism of cancer cells. These data indicate that the presence of Mdm2 at chromatin makes it possible to control the transcription of genes involved in the metabolism and transport of certain amino acids such as serine.

The endogenous serine pool is maintained by a balance between auxotrophy and de novo synthesis, that are strongly deregulated during cell transformation to support the anabolic needs of cancer cells. Mdm2 is recruited via transcription factors of the ATF family on target genes involved in de novo synthesis and serine transport.

Clinicians propose to identify a biological test for the prognosis and diagnosis of LPS that does not require invasive biopsy. Patients included in the study will be patients with WD-LPS or DD-LPS, with the goal of including 100 patients over 2 years.

Based on recent data showing that LPS growth is mediated by Mdm2-mediated regulation of serine metabolism, clinicians propose to measure serine blood levels as a surrogate marker for LPS development. To maintain the intracellular level of serine, Mdm2 controls both de novo serine synthesis (a metabolic pathway that uses the glycolytic intermediate 3-Phospho-Glycerate to generate serine in cells) and the entry of the serine in the cell by auxotrophy. Given the size of LPS, which can often reach several tens of centimeters, clinicians hypothesized that LPS may result in significant demand for serine that could be produced by the microenvironment and transmitted to the tumor by circulating pools of serine and glycine (which can be inter-converted to serine by cells). The profiling of plasma amino acids is of great clinical interest since they are easy to measure by liquid chromatography (HPLC). Clinicians have already validated an HPLC method to measure different amino acids, including serine and glycine, in the serum. Our preliminary data are in line with our hypothesis since the serum serine level is higher in the xenografted mice with patient tumor compared to serum levels measured in the control mice. In addition, in response to treatment with an Mdm2 inhibitor, which induces a drastic reduction in tumor growth, a decrease in circulating serine can be observed.

Clinicians will use an HPLC coupled with mass spectrometry already developed to measure amino acids from Agilent technology. The quantitative analysis of amino acids combines speed and sensitivity with the reliability of the derivation reaction and the analytical technique. These goals are achieved by automated and online derivatization using o-phthalaldehyde (OPA) for primary amino acids and 9-fluorenylmethyl chloroformate (FMOC) for secondary amino acids. Automated derivation is then integrated into robust HPLC analysis. The complete procedure is fast, accurate, sensitive and reproducible using Agilent 1190 HPLC.

The main objective of this project is to identify a new non-invasive biological test for the diagnosis of LPS by measuring circulating serine levels. The current gold standard is the detection of Mdm2 amplification by the FISH.

ELIGIBILITY:
Inclusion Criteria for LPS patients cohort:

Men/women older than 18 years old,

Surgery for :

* Localized WD-LPS and DD-LPS, and/or
* WD-LPS or DD-LPS local relapse, and/or
* WD-LPS or DD-LPS distant relapse and/or
* Deep adipocytic tumor greater than 5 cms, suggestive of atypical lipomatous tumor Patient accepting blood sample, Patient who signed informed consent

Inclusion Criteria for healthy subjects cohort:

Men/women older than 18 years old, Accepting blood sample, Who signed informed consent Matching on sex and age on LPS patient cohort

Exclusion Criteria:

Presence of NeoAdjuvant Treatment for the present cancer, Unaffiliated patient to French Social Protection System, Patient whose follow up is impossible for psychologic, social, geographic, familial reasons Psychiatric illness that would prevent the patient from giving informed consent or being compliant with the study procedures Patient who have another cancer within the 5 years of the inclusion except in situ breast carcinoma, in situ, basocellular carcinoma.

Pregnancy and/or feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2020-08-26 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Sensibility and specificity of circulating serine level for LPS diagnosis | At 3 months post surgery
  Circulating serine level is a quantitative variable evaluated by its concentration

SECONDARY OUTCOMES:
Relapse-free survival (RFS) | Until the study completion: 2 years
  defined as the time measured from the date of surgery treatment to the date of the first documented tumor relapse
Difference in circulating serine level | 18 months after surgery
  Measured between the highest and the lowest rates on pre- and post-surgery blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Nelly FIRMIN, MD, Study Chair — Institut Régional du Cancer de Montpellier (ICM)
Locations (1):
- Institut du Cancer de Montpellier - Val d'Aurelle, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burningham Z, Hashibe M, Spector L, Schiffman JD. The epidemiology of sarcoma. Clin Sarcoma Res. 2012 Oct 4;2(1):14. doi: 10.1186/2045-3329-2-14. PMID 23036164
- [Background] Smolle MA, Tunn PU, Goldenitsch E, Posch F, Szkandera J, Bergovec M, Liegl-Atzwanger B, Leithner A. The Prognostic Impact of Unplanned Excisions in a Cohort of 728 Soft Tissue Sarcoma Patients: A Multicentre Study. Ann Surg Oncol. 2017 Jun;24(6):1596-1605. doi: 10.1245/s10434-017-5776-8. Epub 2017 Jan 20. PMID 28108827
- [Background] Chandrasekar CR, Wafa H, Grimer RJ, Carter SR, Tillman RM, Abudu A. The effect of an unplanned excision of a soft-tissue sarcoma on prognosis. J Bone Joint Surg Br. 2008 Feb;90(2):203-8. doi: 10.1302/0301-620X.90B2.19760. PMID 18256089